CLINICAL TRIAL: NCT05067127
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blinded, Multicenter Study to Evaluate the Efficacy and Safety of Pegcetacoplan in Patients With C3 Glomerulopathy or Immune-Complex Membranoproliferative Glomerulonephritis
Brief Title: Phase III Study Assessing the Efficacy and Safety of Pegcetacoplan in Patients With C3 Glomerulopathy or Immune-Complex Membranoproliferative Glomerulonephritis
Acronym: VALIANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APL2-C3G-310
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: C3G; IC-MPGN; C3 Glomerulopathy; C3 Glomerulonephritis; Complement 3 Glomerulopathy; Complement 3 Glomerulopathy (C3G); Complement 3 Glomerulonephritis; Dense Deposit Disease; DDD; Membranoproliferative Glomerulonephritis; Membranoproliferative Glomerulonephritis (MPGN); Immune Complex Membranoproliferative Glomerulonephritis (IC-MPGN)
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — pegcetacoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Pegcetacoplan administration (Experimental): Subcutaneous infusion of 20mL (1080 mg), twice weekly (for adults or adolescents >50kg), and the three other weight-based doses either of 10mL (540mg), 12mL (648mg), or 15mL (810mg)
  Interventions: Drug: Pegcetacoplan
- Group 2: Placebo administration (Placebo Comparator): Subcutaneous infusion of either 10mL, 12mL, 15mL, or 20mL, twice weekly
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pegcetacoplan — Complement (C3) Inhibitor
  Arms: Group 1: Pegcetacoplan administration
Other: Placebo — Sterile solution of equal volume to active arm
  Arms: Group 2: Placebo administration

SUMMARY:
This is a Phase 3 study to assess the efficacy and safety of twice-weekly subcutaneous (SC) doses of pegcetacoplan compared to placebo in patients with C3 glomerulopathy (C3G) or immune-complex membranoproliferative glomerulonephritis (IC-MPGN) on the basis of a reduction in proteinuria.

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years; where approved, adolescents (aged 12-17 years) weighing at least 30 kg may also be enrolled.
2. A diagnosis of primary C3G or IC-MPGN (with or without previous renal transplant).
3. Evidence of active renal disease, based on one or more of the following:

   1. In adults or adolescents with a baseline renal biopsy (either one collected during screening or a historic biopsy collected within 28 weeks prior to randomization), at least 2+ C3c staining on the baseline renal biopsy.
   2. In adolescents not providing a baseline renal biopsy, at least one of the following:

      * Plasma sC5b-9 level above the upper limit of normal during screening
      * Serum C3 below the LLN during screening
      * Presence of an active urine sediment during screening, as evidenced by hematuria with at least 5 red blood cells (RBCs) per high-power field (HPF) and/or red blood cell casts on local or central microscopic analysis of urine.
      * Presence of C3 nephritic factor within 6 months of screening, based on central laboratory results or medical history.
4. No more than 50% global glomerulosclerosis or interstitial fibrosis on the baseline biopsy for adult participants or adolescent participants providing a baseline biopsy.
5. At least 1 g/day of proteinuria on a screening 24-hour urine collection and a uPCR of at least 1000 mg/g in at least 2 first-morning spot urine samples collected during screening.
6. eGFR ≥30 mL/min/1.73 m2 calculated by the Chronic Kidney Disease-Epidemiology Collaboration creatinine equation for adults or the Bedside Schwartz equation for adolescents.
7. Stable regimen for C3G/IC-MPGN treatment, as described below:

   1. Angiotensin-converting enzyme inhibitor/, angiotensin receptor blocker, and/or sodium-glucose cotransporter-2 inhibitor therapy that is stable and optimized, in the opinion of the investigator, for at least 12 weeks prior to randomization
   2. Stable doses of other medications that can affect proteinuria (eg, steroids, mycophenolate mofetil, and/or other allowed immunosuppressants that the participant is receiving for treatment of C3G or IC-MPGN) for at least 12 weeks prior to the baseline renal biopsy and randomization.
   3. If a participant is on prednisone (or other systemic corticosteroid) for C3G or IC-MPGN treatment, the dosage is stable and no higher than 20 mg/day (or equivalent dosage of a corticosteroid other than prednisone) for at least 12 weeks prior to randomization.
8. Have received vaccinations against S pneumoniae, N meningitidis (types A, C, W, Y, and B), and H influenzae (type B) within 5 years prior to randomization or agree to receive vaccinations during screening.

Exclusion Criteria:

1. Previous exposure to pegcetacoplan.
2. C3G/IC-MPGN secondary to another condition (eg, infection, malignancy, monoclonal gammopathy, a systemic autoimmune disease such as systemic lupus erythematosus, chronic antibody-mediated rejection, or a medication), in the opinion of the investigator.
3. Current or prior diagnosis of human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV) infection or positive serology during screening that is indicative of infection with any of these viruses.
4. Body weight greater than 100 kg at screening.
5. Hypersensitivity to pegcetacoplan or to any of the excipients.
6. History of meningococcal disease.
7. Malignancy, except for the following:

   1. Cured basal or squamous cell skin cancer
   2. Curatively treated in situ disease
   3. Malignancy-free and off treatment for ≥5 years
8. Severe infection (eg, requiring IV antibiotic therapy) within 14 days prior to the first dose of pegcetacoplan.
9. An absolute neutrophil count <1000 cells/mm3 at screening.
10. Use of rituximab, belimumab, or any approved or investigational anticomplement therapy other than pegcetacoplan within 5 half-lives of that product prior to the screening period.
11. Female participants who are pregnant or who are currently breastfeeding and are unwilling to discontinue for the duration of the study and for at least 90 days after the final dose of study drug.
12. Presence or suspicion of severe infection during the screening period (including but not limited to recurrent or chronic infections) that, in the opinion of the investigator, may place the participant at unacceptable risk by study participation.
13. Known or suspected hereditary fructose intolerance.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2025-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (125):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Academic Medical Research Institute, Los Angeles, California
  - Keck School of Medicine, University of Southern California, Los Angeles, California
  - Ronald Reagan UCLA Medical Center (01035), Los Angeles, California
  - UCI Center for Clinical Research, Orange, California
  - UC Davis Medical Center (Transplant Research) (01016), Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Fides Clinical Research, LLC (01042), Atlanta, Georgia
  - Institute for Public Health and Medicine Northwestern University Northwestern University (01041), Chicago, Illinois
  - NANIU Research Chicago (01040), Oak Brook, Illinois
  - Nephrology Associates of Northern IL and Inn (01043), Fort Wayne, Indiana
  - The University of Iowa, Iowa City, Iowa
  - Boston Children's Hospital (01013), Boston, Massachusetts
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Cohen Children Hospital, New Hyde Park, New York
  - CUIMC - Columbia Nephrology, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University (01038), Portland, Oregon
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - MedResearch Inc, El Paso, Texas
  - Texas Children's Hospital, Houston, Texas
- Argentina (3):
  - Hospital Universitario Austral, Buenos Aires
  - Hospital Privado-Universitario de Cordoba, Córdoba
  - Clinica Privada Velez Sarsfield, Córdoba
- Australia (5):
  - Canberra Hospital - Renal Clinical Trials & Research Unit, Garran, Australian Capital Territory
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash University, Box Hill
  - St. Vincents Melbourne, Fitzroy
  - Princess Alexandra Hospital, Woolloongabba
- Austria (2):
  - Medical University Hospital Innsbruck (43004), Innsbruck
  - Medizinische Universität Wien, Vienna
- Belgium (5):
  - Hopital Erasme HUB Service Pharmacie, Brussels
  - University Hospital Antwerp (32004), Edegem
  - Catholic University of Leuven, Leuven
  - CHU Sart-Tilman, Liège
  - Clinical Trials CHU de Liège, Liège
- Brazil (15):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Centro de Tratamento de Doencas Renais, Juiz de Fora, Minas Gerais
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - HC UNESP Botucatu, Botucatu
  - Hospital Universitario Walter Cantidio, Fortaleza
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Real Hospital Portuguas de Beneficancia em Pernambuco, Recife
  - Hospital das Clinicas de Ribeirao Preto, Division of Nephrology, Ribeirão Preto
  - Nefrologia I-Dor, Rio de Janeiro
  - Ruschel Medicina E Pesquisa Clinica, Rio de Janeiro
  - Hospital de Base, São José do Rio Preto
  - UNIFESP - Hospital Sao Paulo, São Paulo
  - Instituto da Crianca-Hospital das Clinicas University of Sao Paulo, São Paulo
  - HCFMUSP-Hospital Clinicas da Faculdade Medicina da Universidade de São Paulo, São Paulo
- Canada (2):
  - Hospital for Sick Children (11003), Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- Czechia (2):
  - Institute for Clinical and Experimental Medicine, Prague
  - Faculty Hospital Kralovske Vinohrady (42002), Prague
- France (11):
  - CHU de Bordeaux - Hopital Pellegrin, Bordeaux
  - Hopital Henri-Mondor, Créteil
  - Hospital Edouard Herriot, Hospices Civils de Lyon, Lyon
  - CHU Montpellier, Hopital Lapeyronie, Montpellier
  - Nantes University Hospital, Nantes
  - Lille Regional University Hospital Center, Claude Huriez Hospital, Department of Nephrology, Paris
  - Hopital Necker (33014), Paris
  - Hôpital Européen Georges-Pompidou, Paris
  - CHU de Saint Etienne, Hospital Nord, Saint-Priest-en-Jarez
  - University Hospital Strasbourg, Strasbourg
  - Rangueil Hospital-University Hospital Center (CHU) of Toulouse, Toulouse
- Germany (6):
  - Charite Universitatsmedizin (49007), Berlin
  - Universitatsklinikum Essen (AoR), Zentrum fur Kinder (49005), Essen
  - Medizinische Hochschule Hannover, Studienzentrum fur Nieren und Hochdruckerkrankungen, Hanover
  - Universitatsmedizin Mainz, Mainz
  - Universitatsklinikum Munster, Münster
  - University Hospital Regensburg (49004), Regensburg
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Institute of Pediatric Nephrology, Petah Tikva
- Italy (9):
  - Policlinico di Bari, Bari
  - Policlinico Sant Orsola-Malpighi, Bologna
  - IRCCS Istituto Giannina Gaslini (39012), Genova
  - Universita degli Studi di Messina, Messina
  - Istituto di Ricerche Farmacologiche Mario Negri IRCCS, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria di Padova (39011), Padua
  - Instituti Clinici Scientifici Maugeri SPA-IRCCS, Pavia
  - Ospedale Pediatrico Bambino Gesu, Rome
- Japan (8):
  - Nagoya University Hospital (81003), Nagoya, Aichi-ken
  - Aichi Children's Health and Medical Center, Ōbu, Aichi-ken
  - Gunma University Hospital (81006), Maebashi, Gunma
  - NHO Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Nagasaki University Hospital (81005), Nagasaki, Nagasaki
  - Seirei Hamamatsu General Hospital (81004), Hamamatsu, Shizuoka
  - Kitano Hospital, Osaka
  - Kyorin University Hospital (81009), Tokyo
- Netherlands (3):
  - Emma Kinderziekenhuis, Amsterdam UMC, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
- Poland (2):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Uniwersytecki Szpital Kliniczny Nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - Yonsei University College of Medicine, Sinchon Severance Hospital, Seoul
  - Seoul National University Hospital (82005), Seoul
  - Seoul National University Hospital, Soeul
- Spain (8):
  - Fundació Puigvert, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Materno-Infantil Vall d' Hebron, Nefrologia Pediatrica, Barcelona
  - Hospital Materno Infantil Sant Joan de Deu, Barcelona
  - Hospital Universitario 12 de Octubre, Nephrology Department, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - University Hospital of Virgen del Rocio, Seville
  - Hospital Universitario Dr Peset, Valencia
- Switzerland (3):
  - Inselspital, Bern University Hospital, Bern
  - CHUV Lausanne, Lausanne
  - Universitatsspital Zurich, Zurich
- United Kingdom (9):
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester
  - University Hospitals of Leicester NHS trust (44003), Leicester
  - Royal Free London NHS Foundation Trust (44015), London
  - Evelina London Children Hospital (44016), London
  - St George'Äôs University Hospitals NHS Foundation Trust (44014), London
  - Imperial College Healthcare NHS Trust, London
  - Great Ormond Street Hospital Foundation Trust, London
  - Royal Manchester Children's Hospital, Manchester
  - Nottingham Children's Hospital, Nottingham

REFERENCES:
- [Derived] Fakhouri F, Bomback AS, Ariceta G, Delmas Y, Dixon BP, Gale DP, Greenbaum LA, Han SH, Isbel N, Le Quintrec M, Licht C, Mastrangelo A, Mizuno M, Neves de Holanda MI, Pickering MC, Remuzzi G, Van De Kar N, Vivarelli M, Walker PD, Wallace D, Zecher D, Francois C, Deschatelets P, Li L, Wang Z, Abad-Franch L, Kinnman N, Lopez-Lazaro L, Szamosi J, Nester CM; VALIANT Trial Investigators Group. Trial of Pegcetacoplan in C3 Glomerulopathy and Immune-Complex MPGN. N Engl J Med. 2025 Dec 4;393(22):2210-2220. doi: 10.1056/NEJMoa2501510. PMID 41337715

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3 randomized, placebo-controlled, double-blinded study was conducted in subjects with complement 3 glomerulopathy (C3G) or primary immune-complex membranoproliferative glomerulonephritis (IC-MPGN) at 122 sites.
Pre-assignment Details: This study consisted of a screening period (10 weeks), 26-week randomized controlled period (RCP), followed by a 26-week open-label period (OLP) and follow-up period (8 weeks). Subjects were randomized to receive pegcetacoplan or placebo in a ratio of 1:1 in RCP. A total of 124 subjects were enrolled in this study.
Groups:
- Randomized Controlled Period: Pegcetacoplan: All adult subjects (regardless of weight) and adolescent subjects with body weight >=50 kilogram (kg) received pegcetacoplan 1080 milligram (mg) subcutaneous (SC) infusion twice weekly for 26 weeks in RCP.
  Adolescent subjects with body weight 35 to <50 kg received pegcetacoplan 648 mg for the first SC infusion and 810 mg SC infusion thereafter twice weekly for 26 weeks in RCP.
  Adolescent subjects with body weight 30 to <35 kg received pegcetacoplan 540 mg for the first 2 SC infusions and 648 mg SC infusion thereafter twice weekly for 26 weeks in RCP.
- Randomized Controlled Period: Placebo: All adult subjects (regardless of weight) and adolescent subjects (with body weight: 30 to <35 kg, 35 to <50 kg, and >=50 kg) received placebo matching with pegcetacoplan SC infusion twice weekly for 26 weeks in RCP.
- Open-Label Period: Pegcetacoplan to Pegcetacoplan: All eligible adult subjects (regardless of weight) and adolescent subjects with body weight >=50 kg who received pegcetacoplan in RCP continued to receive pegcetacoplan 1080 mg SC infusion twice weekly for 26 weeks in OLP.
  Eligible adolescent subjects with body weight 35 to <50 kg who received pegcetacoplan in RCP continued to receive pegcetacoplan 810 mg SC infusion twice weekly for 26 weeks in OLP.
  Eligible adolescent subjects with body weight 30 to <35 kg who received pegcetacoplan in RCP continued to receive pegcetacoplan 648 mg SC infusion twice weekly for 26 weeks in OLP.
- Open-Label Period: Placebo to Pegcetacoplan: All eligible adult subjects (regardless of weight) and adolescent subjects with body weight >=50 kg who received placebo in RCP entered OLP to receive pegcetacoplan 1080 mg SC infusion twice weekly for 26 weeks in OLP.
  Eligible adolescent subjects with body weight 35 to <50 kg who received placebo in RCP entered OLP to receive pegcetacoplan 810 mg SC infusion twice weekly for 26 weeks in OLP.
  Eligible adolescent subjects with body weight 30 to <35 kg who received placebo in RCP entered OLP to receive pegcetacoplan 648 mg SC infusion twice weekly for 26 weeks in OLP.
Period: Randomized Controlled Period (26 weeks)
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo | Open-Label Period: Pegcetacoplan to Pegcetacoplan | Open-Label Period: Placebo to Pegcetacoplan
Started | 63 | 61 | 0 | 0
Completed (Completed RCP and enrolled into OLP.) | 61 | 57 | 0 | 0
Not Completed | 2 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Investigator or Medical Monitor Decision | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Period: Open-Label Period (26 weeks)
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo | Open-Label Period: Pegcetacoplan to Pegcetacoplan | Open-Label Period: Placebo to Pegcetacoplan
Started | 0 (Eligible subjects entered OLP.) | 0 (Eligible subjects entered OLP.) | 61 (Eligible subjects from 'Randomized Controlled Period: Pegcetacoplan' reporting group entered OLP.) | 57 (Eligible subjects from 'Randomized Controlled Period: Placebo' reporting group entered OLP.)
Completed | 0 | 0 | 59 | 55
Not Completed | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Investigator or Medical Monitor Decision | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized subjects.
Groups:
- Randomized Controlled Period: Pegcetacoplan: All adult subjects (regardless of weight) and adolescent subjects with body weight >=50 kg received pegcetacoplan 1080 mg SC infusion twice weekly for 26 weeks in RCP.
  Adolescent subjects with body weight 35 to <50 kg received pegcetacoplan 648 mg for the first SC infusion and 810 mg SC infusion thereafter twice weekly for 26 weeks in RCP.
  Adolescent subjects with body weight 30 to <35 kg received pegcetacoplan 540 mg for the first 2 SC infusions and 648 mg SC infusion thereafter twice weekly for 26 weeks in RCP.
- Total: Total of all reporting groups
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo | Total
Number analyzed (Participants) | 63 | 61 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (17.08) | 23.6 (14.26) | 26.0 (15.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 26 | 28 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian | 9 | 9 | 18
  Black or African American | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 45 | 46 | 91
  Other | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 15 | 10 | 25
  Not Hispanic or Latino | 41 | 47 | 88
  Not Reported | 6 | 2 | 8
  Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Randomized Controlled Period: Change From Baseline in Log-Transformed Urine Protein-to-Creatinine Ratio (uPCR) at Week 26
Description: Baseline uPCR value was calculated as the average of the uPCR measurements from at least 6 of the 9 first-morning spot urine (FMU) samples collected between the start of screening and Day 1, inclusive. The uPCR values used to calculate baseline included those from the samples collected on Day -2, Day -1, and before dosing on Day 1. In situations where less than 6 samples or more than 9 samples were collected, the average of all collected samples was used for baseline derivation. The difference between treatment groups using a composite contrast of equal-weighted average over Weeks 24, 25, and 26 was estimated.
Time Frame: Baseline (Day -70 to Day 1) to Week 26
Population: The ITT analysis set included all randomized subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: log (uPCR)
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 63 | 61
log (uPCR) | -1.114 [-1.380 to -0.848] | 0.029 [-0.090 to 0.148]
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; An mixed-effect model for repeated measures (MMRM) including fixed categorical effect for treatment group, visit, disease type, baseline immunosuppressants use, stratification factors, and the visit-by-treatment group interactions as well as the continuous, fixed covariate of baseline log-transformed uPCR, was utilized to analyze the log-transformed ratio of uPCR at Week 26 compared to baseline; Test type: Superiority; p < 0.0001, MMRM; Difference in least squares (LS) mean = -1.143, 95% CI 2-sided [-1.436 to -0.85]

2. Secondary Outcome: Randomized Controlled Period: Percentage of Subjects Who Achieved the Composite Renal Endpoint at Week 26
Description: Subject who achieved a composite renal endpoint was defined as: (1) a stable or improved estimated glomerular filtration rate (eGFR) compared to baseline (<=15% reduction in eGFR), and (2) a >=50% reduction in uPCR compared to baseline. Percentages are rounded off to the hundredth decimal place.
Time Frame: Week 26
Population: The ITT analysis set included all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 63 | 61
percentage of subjects | 49.21 | 3.28
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; The logistic model included treatment group as independent variable and adjusted for baseline eGFR values, baseline log-transformed uPCR values, disease type, and stratification factors; Test type: Superiority; p < 0.0001, Logistic; Odds Ratio (OR) = 27.516, 95% CI 2-sided [6.105 to 124.026]

3. Secondary Outcome: Randomized Controlled Period: Percentage of Subjects With a Reduction of At Least 50% From Baseline in Urine Protein-to-Creatinine Ratio at Week 26
Description: Baseline uPCR value was calculated as the average of the uPCR measurements from at least 6 of the 9 FMU samples collected between the start of screening and Day 1, inclusive. The uPCR values used to calculate baseline included those from the samples collected on Day -2, Day -1, and before dosing on Day 1. In situations where less than 6 samples or more than 9 samples were collected, the average of all collected samples was used for baseline derivation. Percentages are rounded off to the hundredth decimal place.
Time Frame: Baseline (Day -70 to Day 1) and Week 26
Population: The ITT analysis set included all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 63 | 61
percentage of subjects | 60.32 | 4.92
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; The logistic model included treatment group as independent variable and adjusted for baseline log-transformed uPCR values, disease type, and stratification factors; Test type: Superiority; p < 0.0001, Logistic; Odds Ratio (OR) = 30.932, 95% CI 2-sided [8.401 to 113.897]

4. Secondary Outcome: Randomized Controlled Period: Change From Baseline in the C3 Glomerulopathy (C3G) Histologic Index Activity Score at Week 26
Description: The C3G histologic index used to assess disease activity and chronicity in C3G. The C3G total activity score ranges from 0 (worse) to 21 (best). Higher scores indicate better outcome. Baseline was defined as the most recent non-missing measurement prior to taking the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 26
Population: The ITT analysis set included all randomized subjects. Since adolescents subjects were not required to provide post-screening biopsies, this endpoint was analyzed based on adult subjects only.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 35 | 34
units on a scale | -3.482 [-4.721 to -2.244] | -2.480 [-3.775 to -1.186]
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; Analysis of covariance (ANCOVA) model included treatment as fixed effect, adjusted for baseline C3G histologic index activity score, disease type, and stratification factors; Test type: Superiority; p = 0.2753, ANCOVA; Difference in LS mean = -1.002, 95% CI 2-sided [-2.803 to 0.798]

5. Secondary Outcome: Randomized Controlled Period: Percentage of Subjects Who Showed Decrease in C3c Staining on Renal Biopsy From Baseline at Week 26
Description: Subject who showed decrease in C3c staining was defined as decrease of at least 2 orders of magnitude of intensity from baseline. Percentages are rounded off to the hundredth decimal place.
Time Frame: Baseline (Day 1) and Week 26
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 35 | 34
percentage of subjects | 74.29 | 11.76
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; The logistic model included treatment group as independent variable and adjusted for baseline C3c staining, disease type, and stratification factors; Test type: Superiority; p < 0.0001, Logistic; Odds Ratio (OR) = 27.392, 95% CI 2-sided [6.477 to 115.852]

6. Secondary Outcome: Randomized Controlled Period: Change From Baseline in Estimated Glomerular Filtration Rate at Week 26
Description: Serum samples were collected to determine the eGFR, calculated by using chronic kidney disease-epidemiology collaboration (CKD-EPI) creatinine equation for adults and the Bedside Schwartz equation for adolescents. Baseline eGFR value was calculated using the last non-missing assessment prior to first dose of study drug.
Time Frame: Baseline (Day 1) and Week 26
Population: The ITT analysis set included all randomized subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter (mL)/minute/1.73 m^2
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 63 | 61
milliliter (mL)/minute/1.73 m^2 | -1.497 [-5.892 to 2.899] | -7.808 [-11.570 to -4.047]
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; An MMRM model included fixed categorical effect for treatment group, visit, disease type, stratification factors, and the visit-by-treatment group interactions as well as the continuous, fixed covariate of baseline eGFR, was utilized to analyze the mean change from baseline to Week 26 in eGFR; Test type: Superiority; p = 0.0333, MMRM; Difference in LS mean = 6.312, 95% CI 2-sided [0.501 to 12.122]

7. Secondary Outcome: Randomized Controlled Period: Percentage of Subjects Who Achieved Proteinuria <1 Gram (g)/Day at Week 24
Description: Urine samples were collected to determine the proteinuria. Percentage of subjects who achieved proteinuria <1 g/day was assessed by 24-hour urine protein. Percentages are rounded off to the hundredth decimal place.
Time Frame: Week 24
Population: The ITT analysis set included all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 63 | 61
percentage of subjects | 36.51 | 11.48
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; The logistic model included treatment group as independent variable and adjusted for baseline proteinuria values, disease type, and stratification factors; Test type: Superiority; p = 0.0006, Logistic; Odds Ratio (OR) = 5.753, 95% CI 2-sided [2.106 to 15.716]

8. Secondary Outcome: Randomized Controlled Period: Percentage of Subjects With Normalization of Serum Albumin Levels at Week 26
Description: Baseline serum albumin value was calculated as the average of up to 2 serum albumin measurements preceding and including Day 1. Week 26 serum albumin values was calculated as the average of up to 2 serum albumin measurements preceding and including Week 26, no earlier than Week 20 measurement. Percentages are rounded off to the hundredth decimal place.
Time Frame: Week 26
Population: The ITT analysis set included all randomized subjects. Only subjects with serum albumin levels below lower limit of normal (LLN) at baseline are analyzed.
Measure: Number; unit: percentage of subjects
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 27 | 23
percentage of subjects | 77.78 | 4.35
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; The logistic model included treatment group as independent variable and adjusted for baseline albumin values, disease type, and stratification factors; Test type: Superiority; p = 0.0001, Logistic; Odds Ratio (OR) = 88.341, 95% CI 2-sided [8.863 to 880.544]

9. Secondary Outcome: Randomized Controlled Period: Percentage of Subjects With Serum C3 Levels Above the Lower Limit of Normal at Week 26
Description: Baseline serum C3 value was calculated as the average of up to 2 serum C3 measurements preceding and including Day 1. Week 26 serum C3 value was calculated as the average of up to 2 serum C3 measurements preceding and including Week 26, no earlier than Week 20 measurement. Percentages are rounded off to the hundredth decimal place.
Time Frame: Week 26
Population: The ITT analysis set included all randomized subjects. Only subjects with serum C3 levels below LLN at baseline are analyzed.
Measure: Number; unit: percentage of subjects
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 41 | 49
percentage of subjects | 90.24 | 6.12
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; The logistic model included treatment group as independent variable and adjusted for baseline C3 levels, stratification factors and disease type; Test type: Superiority; p = 0.0094, Logistic; Odds Ratio (OR) = 999.999, 95% CI 2-sided [12.175 to 9999.999]

10. Secondary Outcome: Randomized Controlled Period: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 26
Description: The FACIT-Fatigue scale was a 13-item Likert scaled instrument that was self-administered by subjects. Subjects were presented with 13 statements and asked to indicate their responses as it applied to the past 7 days. The 5 possible responses were "not at all" (0), "a little bit" (1), "somewhat" (2), "quite a bit" (3) and "very much" (4). With 13 statements the total score has a range of 0 (worse health-related quality of life) to 52 (best health-related quality of life). Higher scores indicate better quality of life. Baseline was defined as the most recent non-missing measurement prior to taking the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 26
Population: The ITT analysis set included all randomized subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 63 | 61
units on a scale | 0.929 [-1.549 to 3.407] | 0.367 [-1.949 to 2.683]
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; The ANCOVA model included treatment as fixed effect, adjusted for baseline, disease type, and stratification factors; Test type: Superiority; p = 0.7384, ANCOVA; Difference in LS mean = 0.562, 95% CI 2-sided [-2.739 to 3.863]

11. Secondary Outcome: Randomized Controlled Period: Change From Baseline in the Kidney Disease Quality of Life (KDQOL) Score at Week 26
Description: The KDQOL score was constructed as the KDQOL-36 Summary Score (KSS) by averaging the 24 items from Burden of Kidney Disease, Symptoms and Problems of Kidney Disease, and Effects of Kidney Disease on scale ranging from 0 (worse health-related quality of life) to 100 (best health-related quality of life). Higher scores indicate better quality of life. Baseline was defined as the most recent non-missing measurement prior to taking the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 26
Population: The ITT analysis set included all randomized subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo
Number analyzed (Participants) | 63 | 61
units on a scale | 0.757 [-2.385 to 3.900] | -0.587 [-3.847 to 2.672]
Statistical Analysis 1: Comparison: Randomized Controlled Period: Pegcetacoplan vs Randomized Controlled Period: Placebo; The ANCOVA model included treatment as fixed effect, adjusted for baseline, disease type, and stratification factors; Test type: Superiority; p = 0.5648, ANCOVA; Difference in LS mean = 1.345, 95% CI 2-sided [-3.237 to 5.927]

ADVERSE EVENTS:
Time Frame: TEAE data is reported from first dose of study drug (Day 1) up to 56 days after the last dose of study drug (Week 52), up to 60 weeks. All-cause mortality: From first dose of study drug (Day 1) up to end of the study, approximately 137 weeks.
Description: The safety set included all subjects who received at least 1 dose of study drug.
Arm/Group | Randomized Controlled Period: Pegcetacoplan | Randomized Controlled Period: Placebo | Open-Label Period: Pegcetacoplan to Pegcetacoplan | Open-Label Period: Placebo to Pegcetacoplan
All-Cause Mortality (participants affected / at risk) | 1/63 | 0/61 | 0/61 | 0/57
Serious Adverse Events (participants affected / at risk) | 6/63 | 6/61 | 6/61 | 4/57
Other Adverse Events (participants affected / at risk) | 53/63 | 56/61 | 47/61 | 42/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Controlled Period: Pegcetacoplan (N=63) | Randomized Controlled Period: Placebo (N=61) | Open-Label Period: Pegcetacoplan to Pegcetacoplan (N=61) | Open-Label Period: Placebo to Pegcetacoplan (N=57)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster meningoencephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shunt infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Controlled Period: Pegcetacoplan (N=63) | Randomized Controlled Period: Placebo (N=61) | Open-Label Period: Pegcetacoplan to Pegcetacoplan (N=61) | Open-Label Period: Placebo to Pegcetacoplan (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 5 (5) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 4 (5) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 7 (8) | 4 (5) | 8 (9)
Nausea (Gastrointestinal disorders) | 6 (8) | 4 (4) | 6 (10) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (7) | 9 (13) | 7 (10) | 2 (3)
Asthenia (General disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (2)
Fatigue (General disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Infusion site erythema (General disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (54)
Infusion site pain (General disorders) | 1 (1) | 4 (5) | 0 (0) | 2 (3)
Infusion site swelling (General disorders) | 0 (0) | 1 (2) | 1 (1) | 3 (3)
Injection site pain (General disorders) | 2 (2) | 5 (11) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 2 (33) | 7 (48) | 1 (44) | 4 (22)
Oedema (General disorders) | 3 (4) | 5 (6) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 12 (14) | 7 (7) | 5 (7) | 4 (4)
COVID-19 (Infections and infestations) | 2 (2) | 4 (4) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 3 (4) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (15) | 7 (8) | 7 (9) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5) | 4 (5) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 1 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 6 (6) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 8 (20) | 11 (14) | 4 (7) | 7 (8)
Proteinuria (Renal and urinary disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1) | 4 (5) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (5)
Hypertension (Vascular disorders) | 3 (5) | 5 (5) | 6 (6) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT05067127/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT05067127/SAP_001.pdf